CLINICAL TRIAL: NCT02127320
Title: A Randomized, Open Label Crossover Study to Investigate the Pharmacokinetic Drug Interactions Between Rosuvastatin and Ezetimibe in Healthy Male Subjects
Brief Title: Investigating the Pharmacokinetic Drug Interactions Between Rosuvastatin and Ezetimibe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ROZE-101
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental): Rosuvastatin 20mg → Ezetimibe 10mg → Rosuvastatin 20mg and Ezetimibe 10mg
  Interventions: Drug: Rosuvastatin 20mg; Drug: Ezetimibe 10mg; Drug: Rosuvastatin 20mg + Ezetimibe 10mg
- Sequence 2 (Experimental): Rosuvastatin 20mg and Ezetimibe 10mg→ Rosuvastatin 20mg → Ezetimibe 10mg
  Interventions: Drug: Rosuvastatin 20mg; Drug: Ezetimibe 10mg; Drug: Rosuvastatin 20mg + Ezetimibe 10mg
- Sequence 3 (Experimental): Ezetimibe 10mg → Rosuvastatin 20mg and Ezetimibe 10mg → Rosuvastatin 20mg
  Interventions: Drug: Rosuvastatin 20mg; Drug: Ezetimibe 10mg; Drug: Rosuvastatin 20mg + Ezetimibe 10mg
- Sequence 4 (Experimental): Rosuvastatin 20mg and Ezetimibe 10mg → Ezetimibe 10mg → Rosuvastatin 20mg
  Interventions: Drug: Rosuvastatin 20mg; Drug: Ezetimibe 10mg; Drug: Rosuvastatin 20mg + Ezetimibe 10mg
- Sequence 5 (Experimental): Ezetimibe 10mg → Rosuvastatin 20mg → Rosuvastatin 20mg and Ezetimibe 10mg
  Interventions: Drug: Rosuvastatin 20mg; Drug: Ezetimibe 10mg; Drug: Rosuvastatin 20mg + Ezetimibe 10mg
- Sequence 6 (Experimental): Rosuvastatin 20mg → Rosuvastatin 20mg and Ezetimibe 10mg → Ezetimibe 10mg
  Interventions: Drug: Rosuvastatin 20mg; Drug: Ezetimibe 10mg; Drug: Rosuvastatin 20mg + Ezetimibe 10mg

INTERVENTIONS:
Drug: Rosuvastatin 20mg
Drug: Ezetimibe 10mg
Drug: Rosuvastatin 20mg + Ezetimibe 10mg

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic drug interactions between Rosuvastatin and Ezetimibe in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer, age 19~45 years
* The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 28 kg/m2
* Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial.

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study
* History of relevant drug allergies or clinically significant hypersensitivity reaction.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Rosuvastatin AUCτ,ss | 1D 0h(predose), 9D 0h, 10D 0h, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 11D 0h, 12D 0h, 13D 0h
Rosuvastatin Cmax,ss | 1D 0h(predose), 9D 0h, 10D 0h, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 11D 0h, 12D 0h, 13D 0h
Ezetimibe Cmax,ss | 1D 0h(predose), 9D 0h, 10D 0h, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 11D 0h, 12D 0h, 13D 0h
Ezetimibe AUCτ,ss | 1D 0h(predose), 9D 0h, 10D 0h, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 11D 0h, 12D 0h, 13D 0h

SECONDARY OUTCOMES:
Rosuvastatin Tmax,ss | 1D 0h(predose), 9D 0h, 10D 0h, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 11D 0h, 12D 0h, 13D 0h
Rosuvastatin t1/2β | 1D 0h(predose), 9D 0h, 10D 0h, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 11D 0h, 12D 0h, 13D 0h
Ezetimibe Tmax,ss | 1D 0h(predose), 9D 0h, 10D 0h, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 11D 0h, 12D 0h, 13D 0h
Ezetimibe t1/2β | 1D 0h(predose), 9D 0h, 10D 0h, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 11D 0h, 12D 0h, 13D 0h

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Seok Lim, MD PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Korea, Republic of, South Korea